CLINICAL TRIAL: NCT03569228
Title: Efficacy of a Coupler-based Fitting Approach for Experienced Users Receiving Replacement Hearing Aids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not achieve recruitment goal due to COVID delays and staffing.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2777-R
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aids
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Study 1. Participants obtaining replacement in-the-ear (ITE) or behind-the ear (BTE) hearing aids will be assigned to the ITE or BTE coupler-based fitting groups.
  Study 2: Participants will be fitted with open-fit hearing aids using simulated audiograms.
  Study 3. Participants obtaining replacement open fit or receiver-in-the canal hearing aids will be randomly assigned to the standard of care fitting groups (open or closed) or the coupler-based fitting groups (open or closed).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (7):
- Study 1 (In-the-Ear) Group (Experimental): Experienced users of in-the-ear (ITE) hearing aids will receive replacement ITE hearing aids that are fitted and verified in a test box coupler, then mailed to the patient for a 4-week field trial.
  Interventions: Device: Study 1 - ITE hearing aids
- Study 1 (Behind-the-Ear) Group (Experimental): Experienced users of behind-the-ear (BTE) hearing aids will receive replacement BTE hearing aids that are fitted and verified in a test box coupler, then mailed to the patient for a 4-week field trial.
  Interventions: Device: Study 1 - BTE hearing aids
- Study 2 (Open-Fit corrections) (No Intervention): Participants with hearing loss will be fitted monaurally with 12 stock non-custom, receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids using the standard in-situ approach and test box measures will be made of each fitting to develop correction factors for these styles.
- Study 3 (open-fit comparison) (Active Comparator): This group will serve as the active comparator group for experienced hearing aid user receiving replacement receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids with OPEN coupling using the standard of care approach, then undergoing a 4-week field trial.
  Interventions: Device: Study 3 (open-fit comparison)
- Study 3 (closed-fit comparison) (Active Comparator): This group will serve as the active comparator group for experienced hearing aid user receiving replacement receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids with CLOSED coupling using the standard of care approach, then undergoing a 4-week field trial.
  Interventions: Device: Study 3 (closed-fit comparison)
- Study 3 (experimental open-fit) (Experimental): Experienced hearing aid user receiving replacement receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids with OPEN coupling that are fitted and verified in a test box coupler, then mailed to the patient for a 4-week field trial.
  Interventions: Device: Study 3 (experimental open-fit)
- Study 3 (experimental closed-fit) (Experimental): Experienced hearing aid user receiving replacement receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids with CLOSED coupling that are fitted and verified in a test box coupler, then mailed to the patient for a 4-week field trial.
  Interventions: Device: Study 3 (experimental closed-fit)

INTERVENTIONS:
Device: Study 1 - ITE hearing aids — Experienced users of in-the-ear (ITE) hearing aids will receive replacement ITE hearing aids that are fitted and verified in a test box coupler, then mailed to the patient for a 4-week field trial.
  Arms: Study 1 (In-the-Ear) Group
Device: Study 1 - BTE hearing aids — Experienced users of behind-the-ear (BTE) hearing aids will receive replacement BTE hearing aids that are fitted and verified in a test box coupler, then mailed to the patient for a 4-week field trial.
  Arms: Study 1 (Behind-the-Ear) Group
Device: Study 3 (open-fit comparison) — This group will serve as the active comparator group for experienced hearing aid user receiving replacement receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids with OPEN coupling using the standard of care approach, then undergoing a 4-week field trial.
  Arms: Study 3 (open-fit comparison)
Device: Study 3 (closed-fit comparison) — This group will serve as the active comparator group for experienced hearing aid user receiving replacement receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids with CLOSED coupling using the standard of care approach, then undergoing a 4-week field trial.
  Arms: Study 3 (closed-fit comparison)
Device: Study 3 (experimental open-fit) — Experienced hearing aid user receiving replacement receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids with OPEN coupling that are fitted and verified in a test box coupler, then mailed to the patient for a 4-week field trial.
  Arms: Study 3 (experimental open-fit)
Device: Study 3 (experimental closed-fit) — Experienced hearing aid user receiving replacement receiver in the canal (RIC) or receiver in the aid (RITA) hearing aids with CLOSED coupling that are fitted and verified in a test box coupler, then mailed to the patient for a 4-week field trial.
  Arms: Study 3 (experimental closed-fit)

SUMMARY:
Hearing loss is among the top service-connected disabilities in Veterans. Hearing aids are the primary intervention for hearing loss. Half of the hearing aids dispensed in the VA are to Veterans who are receiving replacement amplification. Many Veterans would like their replacement hearing aids mailed to them, but they are required to travel to the clinic so that the fit of the hearing aid can be verified. There are standard fitting procedures, such as those used in infants and children, that use a coupler to simulate the patient's real ear to verify the hearing aid fitting. The results of this study should determine the efficacy of a coupler-based hearing-aid fitting protocol that would not require the Veteran to attend the fitting appointment, thereby contributing to improved Veteran-Centric care.

DETAILED DESCRIPTION:
In the VA system, hearing loss is the second-most common service-connected condition affecting 933,182 Veterans, exceeded only by tinnitus which affects 1,121,709 Veterans (data from Veterans Benefit Report for Fiscal Year 2016). In FY 2016, the VA dispensed 750,075 hearing aids at a net procurement of nearly $270 million (report generated from VA Denver Acquisition and Logistics Center [DALC] Remote Order Entry System [ROES]). Half of the hearing aids dispensed were to experienced hearing aid users receiving replacement hearing aids (Dennis, 2014). VA Audiology caseload is significant and Veterans can experience long wait-times for fitting appointments to obtain new hearing aids (Office of the Inspector General, 2014).

The purpose of the fitting appointment is to program and verify the hearing aids and orient the patient to hearing aid use/care. For patients obtaining replacement hearing aids, the orientation typically is unnecessary, and the programming is simplified; consisting mainly of matching the individual's real-ear aided response (REAR) and hearing aid output to appropriate target values. In contrast to adults, REAR measurements are not well-tolerated by children due to the requirement for placement of a probe tube in the ear canal. Therefore, a hearing aid fitting procedure that circumvents the need for in situ REAR measurements (real ear coupler difference or RECD) is the standard-of-care (SoC) for children. Considerable research clearly has shown the equivalency of in situ REAR and RECD fitting procedures (e.g., Moodie et al., 1994). RECD fitting procedures rarely are used with adults; however, such an approach could preclude the need for direct physical contact with the patient at the time of the hearing aid fitting. Three experiments are proposed. The purpose of the first study is to evaluate coupler-based fitting approach for groups of experienced users obtaining replacement hearing aids and compare the accuracy of those fittings to the prescription and their outcomes to norms. The second study aims to develop correction factors for venting of open-fit hearing aids. The third study will focus on comparing coupler-based fittings of open-fit hearing aids (using correction factors developed from study two results) to an SoC (active control) group who will have their open-fit hearing aids fitted in face-to-face appointment via standard in situ REAR procedures. In Study 1 and 3, both groups will return for in situ REARs and self-report outcomes assessment one month after the hearing-aid fitting. The results of this study should determine the efficacy of a RECD-based, hearing-aid fitting approach for experienced hearing-aid users who are receiving replacement hearing aids consisting of a variety of styles. If the approaches are equivalent, then this study will provide an evidence-based, RECD fitting approach that should result in greater patient satisfaction and reduced costs.

ELIGIBILITY:
Inclusion Criteria:

Study 1 and 3

* experienced hearing-aid users who are obtaining replacement VA-issued hearing aids of the same style and manufacturer as their current hearing aids
* no more than a moderate sensorineural hearing loss (defined as < 60 dB HL pure-tone average at 500, 1000, and 2000 Hz AU)
* symmetrical hearing between the ears as defined as no more than a 20 dB difference in pure-tone thresholds at two consecutive frequencies
* 50% word-recognition abilities in quiet as measured during the diagnostic audiologic evaluation
* An education-adjusted score of >21 on the Montreal Cognitive Assessment
* ability to read and write in English

Study 2 Veterans aged 18-85 years with sensorineural hearing loss

Exclusion Criteria:

Study 1 and 3

* outer or middle ear pathology as determined by otoscopy, immittance, and/or audiometric testing (e.g., conductive or mixed losses)
* a significant change in hearing on audiogram obtained during the current study and that obtained when fitted with the current (to-be replaced) hearing aids as defined by a 15 dB decline in thresholds at three consecutive frequencies in either ear
* lack of phone or non-use of the phone
* unwilling or unable to be mailed hearing aids
* co-morbid condition that would preclude their participation

Study 2

* co-morbid condition that would preclude their participation
* outer or middle ear pathology as determined by otoscopy, immittance, and/or audiometric testing (e.g., conductive or mixed losses)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candice M Quinn, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded from the study only if they failed pre-screening.
  In Study 2, participants were randomly assigned a sham audiogram. Participants in Study 2 were fit with 12 hearing aids and the "outcome" was deviation to target. Study 2 participants do not have the same pre-specified primary and secondary outcomes as those in Study 1 and 3 and not reported.
Groups:
- Study 2 (Open Fit Correction, Sham Audiogram 1): Sham Audiogram 1 represents a normal sloping to moderate sensorineural hearing loss. Please note: participants in this arm did not have this audiogram.
- Study 2 (Open Fit Correction, Sham Audiogram 2): Sham Audiogram 2 represents a gradual normal sloping to moderate sensorineural hearing loss in participants. Please note: participants did not have this audiogram.
- Study 2 (Open Fit Correction, Sham Audiogram 3): Sham Audiogram 3 represents a mild to severe sensorineural hearing loss. Please note: participants did not have this audiogram.
Period: Overall Study
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 2 (Open Fit Correction, Sham Audiogram 1) | Study 2 (Open Fit Correction, Sham Audiogram 2) | Study 2 (Open Fit Correction, Sham Audiogram 3) | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit)
Started | 4 | 11 | 35 | 37 | 32 | 12 | 9 | 14 | 9
Completed | 2 | 9 | 32 | 34 | 30 | 9 | 8 | 9 | 6
Not Completed | 2 | 2 | 3 | 3 | 2 | 3 | 1 | 5 | 3
Not completed — Withdrawal by PI | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Screen Fail | 2 | 2 | 1 | 1 | 1 | 3 | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Study 2 (Open-fit Corrections, Sham Audiogram 1): Sham Audiogram 1 represents normal sloping to moderate sensorineural hearing loss.
- Study 2 (Open-fit Corrections, Sham Audiogram 2): Sham Audiogram 2 represents gradual normal sloping to moderate sensorineural hearing loss.
- Study 2 (Open-fit Corrections, Sham Audiogram 3): Sham Audiogram 3 represents mild sloping to severe sensorineural hearing loss.
- Total: Total of all reporting groups
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 2 (Open-fit Corrections, Sham Audiogram 1) | Study 2 (Open-fit Corrections, Sham Audiogram 2) | Study 2 (Open-fit Corrections, Sham Audiogram 3) | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit) | Total
Number analyzed (Participants) | 2 | 9 | 32 | 34 | 30 | 9 | 8 | 9 | 6 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (6.4) | 75.6 (4.4) | 72.5 (6.8) | 72.6 (6.9) | 74.7 (5.0) | 73.2 (6.6) | 74.3 (4.6) | 69.1 (10.5) | 74.8 (4.8) | 73.3 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Male | 2 | 9 | 31 | 33 | 30 | 9 | 8 | 9 | 6 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 9 | 32 | 34 | 30 | 8 | 8 | 9 | 6 | 138
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 4 | 2 | 0 | 0 | 3 | 0 | 10
  White | 1 | 8 | 31 | 28 | 28 | 9 | 8 | 6 | 6 | 125
  More than one race | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 9 | 32 | 34 | 30 | 9 | 8 | 9 | 6 | 139

OUTCOME MEASURES:

1. Primary Outcome: Deviation From Target (in dB)
Description: The primary outcome of interest is based on fitting accuracy across ears (i.e., the averaged absolute deviation from target of the average of 500, 1000, 2000, and 4000 Hz across both ears measured in decibels (dB)).
Time Frame: 1 month
Population: Only groups in Studies 1 and 3 are included. Study 2 is a single session observational study to determine correction factors for Study 3. Study 2 is not included for this purpose.
Measure: Mean (Standard Deviation); unit: units on a scale (dB)
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit)
Number analyzed (Participants) | 2 | 9 | 9 | 8 | 9 | 6
units on a scale (dB) | 0 (0) | 2.85 (2.69) | 6.5 (6.7) | 6.6 (5.8) | 4.6 (4.9) | 3.5 (4.8)

2. Secondary Outcome: Abbreviate Profile of Hearing Aid Benefit
Description: Abbreviate Profile of Hearing Aid Benefit (APHAB; Cox and Alexander, 1995). The APHAB contains 24 items that assess hearing problems across four subscales including: (1) ease of communication, (2) background noise, (3) reverberation, and (4) aversiveness to sounds. Items are answered using a 7-item response scale ranging from never (1%) to almost always (99%). Items typically are answered in unaided and aided conditions. Higher numbers indicated more problems. The difference in scores between the two conditions is a measure of benefit. For this study, however, the aided-aided version of the APHAB will be used. Study 1 and 3.
Time Frame: 1 month
Population: Only groups in Studies 1 and 3 are included. In the Study 3 closed-fit comparison group, 2 had missing APHAB outcomes. Study 2 is a single session observational study to determine correction factors for Study 3. Study 2 is not included for this purpose.
Measure: Mean (Standard Deviation); unit: units on a 1 to 99 percent scale
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit)
Number analyzed (Participants) | 2 | 9 | 9 | 6 | 9 | 6
units on a 1 to 99 percent scale | 12.1 (1.6) | 25.1 (13.5) | 29.1 (13.8) | 18.8 (10.4) | 26.9 (12.6) | 21.3 (12.0)

3. Secondary Outcome: Client-Oriented Scale of Improvement
Description: Client-Oriented Scale of Improvement (COSI; Dillon, James, & Ginis, 1997). The listener nominates up to five listening goals on the COSI. After hearing-aid use, the listener assesses two outcomes for each goal. One outcome is the "degree of change" relative to the patient's unaided experience. Responses are recorded on a categorical scale from 'worse' to 'much better.' The second outcome is the final satisfactory "aided" ability for each goal as measured on a categorical scale from hardy ever (10%) to almost always (95%). The percentage of 'better' and 'much better' responses and the average of the final ability will be calculated across goals. Study 1 and 3.
Time Frame: 1 month
Population: Only groups in Studies 1 and 3 are included. Study 2 is a single session observational study to determine correction factors for Study 3. Study 2 is not included for this purpose. Study 2 participants were not administered patient reported outcome measures nor did they undergo a field trial with hearing aids.
Measure: Mean (Standard Deviation); unit: percentage of final ability
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit)
Number analyzed (Participants) | 2 | 9 | 9 | 8 | 9 | 6
percentage of final ability | 61.7 (16.5) | 71.6 (19.3) | 71.8 (20.3) | 77.6 (18.5) | 72.7 (22.8) | 67.5 (22.0)

4. Secondary Outcome: International Outcomes Inventory for Hearing Aids
Description: International Outcomes Inventory for Hearing Aids (IOI-HA; Cox et al., 2000). The IOI-HA consists of seven items including (1) use, (2) benefit, (3) satisfaction, (4) residual activity limitation, (5) residual participation restriction, (6) impact on others, and (7) quality of life. Each item has a unique 1-5 response scale. Scores range from 7-35 with higher scores indicating higher outcomes. Study 1 and 3.
Time Frame: 1 month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a 1 to 5 scale, summed
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit)
Number analyzed (Participants) | 2 | 9 | 9 | 8 | 9 | 6
units on a 1 to 5 scale, summed | 31.0 (1.4) | 30.4 (3.0) | 30.9 (2.5) | 31.0 (4.0) | 28.8 (3.5) | 30.5 (2.6)

5. Secondary Outcome: Satisfaction With Amplification in Daily Life
Description: Satisfaction with Amplification in Daily Life (SADL) (Cox and Alexander, 1999). The SADL questionnaire has 15 items that examine self-reported hearing-aid satisfaction. The following four subscales are included: (1) positive effect, (2) negative features, (3) personal image, and (4) service and cost. For the current study, item 14 on the service and cost subscale will not be used as the Veterans are not charged for the cost of their bilateral hearing aids. The SADL uses a 7-item response scale in 1-unit steps, 1 (poorest) to 7 (highest) for each item, which are averaged for each subscale and total scale score. Study 1 and 3.
Time Frame: 1 month
Population: In the Study 3 closed-fit comparison group, 2 had missing SADL outcomes. Study 2 did not include outcome measures as it was not a clinical trial. Study 2 was a one-session observational study required to develop corrections for Study 3.
Measure: Mean (Standard Deviation); unit: units on a 1 to 7 scale
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit)
Number analyzed (Participants) | 2 | 9 | 9 | 6 | 9 | 6
units on a 1 to 7 scale | 6.1 (0.5) | 6.1 (0.4) | 5.8 (0.8) | 6.5 (0.2) | 6.0 (0.5) | 6.3 (0.3)

6. Secondary Outcome: Client Oriented Scale of Improvement (COSI)
Description: Degree of change (percentage of those goals that were categorized as 'better' or 'much better')
Time Frame: 1 month
Population: Only groups in Studies 1 and 3 are included. In the Study 3 closed-fit comparison group, 2 had missing COSI outcomes. Study 2 is a single session observational study to determine correction factors for Study 3. Study 2 is not included for this purpose. Study 2 participants were not administered patient reported outcome measures nor did they undergo a field trial with hearing aids.
Measure: Number; unit: percentage of 'better' or 'much better'
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit)
Number analyzed (Participants) | 2 | 9 | 9 | 6 | 9 | 6
percentage of 'better' or 'much better' | 25 | 56.25 | 62 | 87.5 | 51.8 | 25

7. Other Pre Specified Outcome: Deviation From Target for Open-Fit Corrections
Description: Deviation from target (dB) averaged from 500 - 4000Hz across all 12 sham fittings. This is the sole outcome measure for Study 2 participants only. Study 1 and Study 3 participants do not have this outcome measure.
Time Frame: Single session laboratory-based observational visit
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Study 2 (Open Fit Correction, Sham Audiogram 1) | Study 2 (Open Fit Correction, Sham Audiogram 2) | Study 2 (Open Fit Correction, Sham Audiogram 3)
Number analyzed (Participants) | 32 | 34 | 30
dB | 0.95 (2.21) | 1.98 (3.52) | 4.54 (3.21)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Study 1 (In-the-Ear) Group | Study 1 (Behind-the-Ear) Group | Study 2 (Open-Fit Corrections, Sham Audiogram 1) | Study 2 (Open-Fit Corrections, Sham Audiogram 2) | Study 2 (Open-Fit Corrections, Sham Audiogram 3) | Study 3 (Open-fit Comparison) | Study 3 (Closed-fit Comparison) | Study 3 (Experimental Open-fit) | Study 3 (Experimental Closed-fit)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/11 | 0/32 | 0/34 | 0/30 | 0/12 | 0/9 | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/11 | 0/32 | 0/34 | 0/30 | 0/12 | 0/9 | 0/14 | 0/9
Other Adverse Events (participants affected / at risk) | 0/4 | 0/11 | 0/32 | 0/34 | 0/30 | 0/12 | 0/9 | 0/14 | 0/9

LIMITATIONS AND CAVEATS:
Early termination due to small number of subjects analyzed. Study 2 was not a clinical trial and data used to inform correction factors for Study 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03569228/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT03569228/ICF_001.pdf